CLINICAL TRIAL: NCT06428331
Title: A Phase 1, Multicenter, Open-label First-In-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antitumor Activity of SKB518 in Subjects With Advanced Solid Tumors
Brief Title: A Study of SKB518 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB518-I-01
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Several dose levels are tentatively planned for Phase 1
  Interventions: Drug: SKB518 for injection

INTERVENTIONS:
Drug: SKB518 for injection — SKB518 for injection is administered every 3 weeks (q3w) until radiographic disease progression (PD), intolerable toxicity, death, or discontinuation of treatment, whichever occurs first.
  Other Names: SKB518

SUMMARY:
This is a first-in-human (FIH), phase 1, multicenter, open-label, dose-escalation study of SKB518 to evaluate the safety, tolerability, PK, immunogenicity, and antitumor activity in adult subjects with advanced or metastatic solid tumor relapsed/refractory to standard therapies or for which no effective standard therapy is available.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), phase 1, multicenter, open-label, dose-escalation study of SKB518 to evaluate the safety, tolerability, PK, immunogenicity, and antitumor activity in adult subjects with advanced or metastatic solid tumor relapsed/refractory to standard therapies or for which no effective standard therapy is available. Dose escalation and de-escalation decisions are based on the mTPI-2 design and depend on the number of subjects enrolled and the number of DLTs observed at the current dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age at the time of signing the informed consent;
2. Histological or cytological diagnosis of solid tumor that is advanced/metastatic solid tumor by pathology report and have progressed on, have been intolerant to, or have been ineligible for standard of care treatments.
3. Subjects able to provide tumor blocks or 8~10 slides [fresh paraffin-embedded tumor tissue or archived paraffin-embedded tumor tissue (maximum time limit is not more than 2 years)] before the first dose of study intervention for biomarkers testing.
4. At least one measurable lesion can be accurately measured per RECIST v1.1 as determined by the local site investigator/radiology assessment. Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
5. Subjects with Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
6. Life expectancy of at least 3 months as assessed by the investigators.
7. Subjects with adequate organ and bone marrow function confirmed by laboratory results within 7 days prior to the first dose.
8. Has recovered from all toxicities from previous therapy with the exception of stable, chronic (>3 months) toxicities not considered a safety risk (e.g. alopecia, vitiligo), after consultation with the Sponsor.
9. Subjects of childbearing potential (male or female) must use effective medical contraception during the study until 6 months after the last dose.
10. Subjects must be able to provide documented voluntary informed consent.

Exclusion Criteria:

1. Has known active or untreated central nervous system (CNS) metastases and/or carcinomatous meningitis are not eligible.
2. Has a known additional malignancy that is progressing or has required active treatment within the past 5 years.
3. Has a history of major cardiovascular, cerebrovascular or thromboembolic diseases.
4. Has serious and/or uncontrolled concomitant diseases.
5. Has known active tuberculosis.
6. Has known human immunodeficiency virus (HIV) infection that is not well controlled.
7. Has any active viral hepatitis, hepatitis B or hepatitis C.
8. Has had major surgery within 28 days prior to the first dose.
9. Has known allergy or hypersensitivity to SKB518, or the excipients of SKB518.
10. Has a history of interstitial lung disease (ILD) or a history of non-infectious pneumonitis that required steroids.
11. Clinically serious lung injuries caused by lung diseases.
12. History of documented severe dry eye syndrome.
13. Has a history of allogeneic tissue/solid organ transplant.
14. Has known uncontrollable effusion.
15. Subjects who are vaccinated with live vaccine within 30 days before the first dose, or plan to be vaccinated with live vaccine during the study period.
16. Has received strong cytochrome P450 (CYP3A4) inhibitors or inducers, or has received BCRP inhibitors within 2 weeks prior to the first dose.
17. Subjects who received any chemotherapy, radiotherapy, immunotherapy, or biologic therapy treatment within 4 weeks; or who received any small molecular tyrosine kinase inhibitor, antitumor hormonal therapy, system immune-stimulator, or therapy with traditional Chinese medicines approved for antitumor treatment, etc. within 2 weeks before the first dose.
18. Has an active infection requiring systemic therapy.
19. Subjects with the disease that requires systemic corticosteroid therapy (prednisolone or equivalent dose of similar drugs at a dose of >10 mg/d) or other immunosuppressive therapy within 14 days before the first dose.
20. Is currently participating and receiving study therapy in a study of an investigational agent or has participated and received study therapy in a study of an investigational agent or has used an investigational device within 28 days of fist dose.
21. Before the first dose, the subject's condition deteriorates rapidly.
22. Has a known psychiatric or substance abuse disorders.
23. The Investigator considers other situations that will interfere with the evaluation of the study intervention or the safety of the subjects or the interpretation of the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects achieving Dose-limiting toxicity (DLT) | From data of initial dose until up to 21 days for treatment
  DLT is defined as an adverse event (AE) that meets protocol defined DLT criteria during cycle 1 and is at least possibly related to study drug.
Maximum Tolerated Dose (MTD) | From data of initial dose until up to 21 days for treatment
  Once the dose escalation stopping criteria are met, the MTD estimated by mTPI-2 will be the dose at which the probability of posterior mean of the DLT rate is between 25% and 35%, closest to 30%, and no more than 35%.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months
  The sum of the number of cases with Complete Response (CR) and Partial Response (PR) in all treated tumor patients (CR + PR) divided by the total number of cases.
Progression Free Survival (PFS) | Up to 24 months
  Time from start of treatment to progression of disease (PD) or death, whichever occurs first, in patients with tumors.
Duration of Response (DOR) | Up to 24 months
  Time from the start of the first assessment of CR or PR in tumor patients to PD or death due to any reason.
Overall Survival (OS) | Up to 24 months
  Time from start of treatment to death due to any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Study Chair — Fudan University; Xiaohua Wu, Study Chair — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China, China